CLINICAL TRIAL: NCT04185272
Title: Role of Butyrophilins in Colon Cancers Aggressiveness Evaluation
Brief Title: Butyrophilins Role in Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IMMUNOCOL-IPC 2019-018
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Colonic Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: colon cancer patients and metastatic colon cancer patients will be included in this study. We expect that BTNL molecules expression is different depending of the aggressiveness of the illness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-metastatic colon cancer (Experimental)
  Interventions: Biological: analysis of BTN and BTNL status
- metastatic colon cancer (Experimental)
  Interventions: Biological: analysis of BTN and BTNL status

INTERVENTIONS:
Biological: analysis of BTN and BTNL status — analysis of BTN and BTNL expression in colon cancer and hepatic metastasis

SUMMARY:
quantification of BTNL molecules in colon cancer in order to determinate if their could be used as a prognostic marquer

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years old,
* Signed participation consent,
* Non-metastatic colon cancer immediately resectable or metastatic and liver synchronous for which it was decided a combined colic and liver surgery (metastatic patient at the outset) in multidisciplinary consultation meeting.
* Performance Status (PS) 0 or 1
* affiliated to the social security or beneficiary

Exclusion Criteria:

* Rectal cancer, colon cancer recurrence
* Emergency of colon cancer Surgery
* History of inflammatory disease of the digestive tract (Crohn's disease or ulcerative colitis)
* Patient who received neoadjuvant therapy other than chemotherapy
* Patient treated with immune-suppressors or long-course corticosteroids <12 months
* Pregnant women or likely to be pregnant (without effective contraception) or breastfeeding,
* Person in urgent situation, person under legal protection measure, or unable to express his / her consent,
* Impossibility of submitting to the medical examination of the test for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
evaluation of BTNL3, BTNL8 and BTNL9 expression by transcriptomics and immunohistochemistry | 8 years
  healthy and cancerous colon ad metastasis (if applicable) will be analysed by

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No